CLINICAL TRIAL: NCT06920004
Title: A Phase 3, Randomized, Double-Blinded, Double-Dummy Study Evaluating the Efficacy and Safety of Intravenous Empasiprubart Versus Intravenous Immunoglobulin in Adults With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: A Study to Assess Efficacy and Safety of Empasiprubart Versus IVIg in Adults With CIDP
Acronym: emvigorate
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-117-2401; 2024-520097-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; CIDP; CIDP - Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - empasiprubart + IVIg-placebo (Experimental): During Part A, participants receive empasiprubart and a placebo resembling the IVIg treatment in this arm.
  Interventions: Biological: empasiprubart; Other: IVIg-placebo
- Part A - IVIg + empasiprubart-placebo (Active Comparator): During Part A, participants receive IVIg and a placebo resembling the empasiprubart treatment in this arm.
  Interventions: Biological: IVIg; Other: empasiprubart-placebo
- Part B - empasiprubart (Experimental): After completion of part A, participants can proceed to part B where they receive empasiprubart (no IVIg). Participants from the empasiprubart + IVIg- placebo arm in Part A will receive empasiprubart placebo once to maintain the blind of Part A.
  Interventions: Biological: empasiprubart; Other: empasiprubart-placebo

INTERVENTIONS:
Biological: empasiprubart — Intravenous infusion of empasiprubart
  Arms: Part A - empasiprubart + IVIg-placebo; Part B - empasiprubart
Biological: IVIg — Intravenous infusion of IVIg
  Arms: Part A - IVIg + empasiprubart-placebo
Other: empasiprubart-placebo — A placebo resembling the empasiprubart treatment
  Arms: Part A - IVIg + empasiprubart-placebo; Part B - empasiprubart
Other: IVIg-placebo — A placebo resembling the IVIg treatment
  Arms: Part A - empasiprubart + IVIg-placebo

SUMMARY:
The main purpose of this study is to compare empasiprubart and IVIg for treating people with CIDP. This study consists of a Part A where participants will either receive empasiprubart and a placebo resembling IVIg, or IVIg and a placebo resembling empasiprubart for 24 weeks (6 months). Following Part A, participants will enter Part B in which all participants will receive empasiprubart for 96 weeks (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for CIDP based on EAN/PNS Task Force CIDP guidelines, second revision (2021)
* Has either typical CIDP or 1 of the following CIDP variants: motor CIDP, multifocal CIDP (also known as Lewis-Sumner syndrome), focal CIDP, or distal CIDP
* Has responded to IVIg in the past 5 years
* Receiving treatment with IVIg within a standard optimal maintenance dosing regimen, with a minimum weekly IVIg dose of at least 0.125 g/kg
* Has residual disability and active disease

Exclusion Criteria:

* Besides the indication under study, known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of CIDP or puts the participant at undue risk, including polyneuropathy of other causes
* Meets the criteria for possible or sensory CIDP based on EAN/PNS Task Force CIDP guidelines, second revision (2021)
* Use of other long-acting immunomodulatory treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of ≥1 point compared with baseline in aINCAT score at week 24 | up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).

SECONDARY OUTCOMES:
Change from baseline in I-RODS centile points score at week 24 | up to 24 weeks
  Inflammatory Rasch-built Overall Disability Scale (I-RODS) assesses the limitations of activities and social participation in patients with inflammatory neuropathies like CIDP. The score ranges from 0 to 100 (higher score, worse outcome).
Change from baseline in MRC-SS at week 24 | up to 24 weeks
  The Medical Research Council Sum Score evaluates motor strength. Evaluated on 6 muscle groups on each side, the score varies from 0 to 60 (lower score, worse outcome).
Change from baseline in grip strength (3-day moving average) in the dominant hand at week 24 | up to 24 weeks
  The grip strength will be measured daily by using a Martin-Vigorimeter. The 3 daily measurements of grip strength from the left hand and the 3 daily measurements of grip strength from the right hand will be recorded, and the daily average for the left hand and right hand will be calculated, respectively. The 3-day moving average will be generated based on the average of the obtained averages for each hand on the target day and the preceding 2 days.
Time to reduction of ≥1 point from baseline in aINCAT score | up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in TUG at week 24 | up to 24 weeks
  The Timed Up and Go Test (TUG) is a simple test to assess a person's mobility in which the time expended to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down is measured.
Time to increase of ≥1 point compared with baseline in aINCAT score | Up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in grip strength (3-day moving average) of both hands over time | up to 24 weeks + 96 weeks (Part B)
  The grip strength will be measured daily by using a Martin-Vigorimeter. The 3 daily measurements of grip strength from the left hand and the 3 daily measurements of grip strength from the right hand will be recorded, and the daily average for the left hand and right hand will be calculated, respectively. The 3-day moving average will be generated based on the average of the obtained averages for each hand on the target day and the preceding 2 days.
Change from baseline in grip strength (daily average) for both hands | up to 24 weeks + 96 weeks (Part B)
  The grip strength will be measured daily by using a Martin-Vigorimeter. The 3 daily measurements of grip strength from the left hand and the 3 daily measurements of grip strength from the right hand will be recorded, and the daily average for the left hand and right hand will be calculated, respectively. A daily average will be generated based on the average of the obtained averages for each hand.
Change from baseline in MRC-SS over time | up to 96 weeks (Part B)
  The Medical Research Council Sum Score evaluates motor strength. Evaluated on 6 muscle groups on each side, the score varies from 0 to 60 (lower score, worse outcome).
Change from baseline in aINCAT over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in EQ-5D-5L over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome).
Change from baseline in RT-FSS over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  Rasch-Transformed Fatigue Severity Scale (RT-FSS) is a patient-reported outcome measure to distinguish fatigue from clinical depression.
Change from baseline in SF-12 over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  12-Item Short Form Health Survey (SF-12) is a general patient-reported outcome measure.
Change from baseline in BPI-SF over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  The Brief Pain Inventory-Short Form (BPI-SF) is a patient-reported outcome measure to assess pain severity and pain interference.
PGI-S values over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  The Patient Global Impression of Severity (PGI-S) is a patient-reported outcome measure that reflects the patient's belief about the severity of the illness.
PGI-C values over time | up to 24 weeks (Part A) + 96 weeks (Part B)
  The Patient Global Impression of Change (PGI-C) is a patient- reported outcome measure that reflects the patient's belief about the efficacy of treatment.
Values for work-related and household chore activities of the HRPQ | up to 24 weeks
  The Health-Related Productivity Questionnaire (HRPQ) assesses health-related and work-related productivity, with questions related to 'hours lost because of absenteeism'.
Percentage of scheduled hours lost in total (absenteeism+ presenteeism) | up to 24 weeks
Change from baseline in I-RODS centile points score over time | Up to 96 weeks (Part B)
  Inflammatory Rasch-built Overall Disability Scale (I-RODS) assesses the limitations of activities and social participation in patients with inflammatory neuropathies like CIDP. The score ranges from 0 to 100 (higher score, worse outcome).
Change from baseline in TUG over time | Up to 96 weeks (Part B)
  The Timed Up and Go Test (TUG) is a simple test to assess a person's mobility in which the time expended to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down is measured.
Incidence of antidrug antibodies against empasiprubart in serum | up to 24 weeks (Part A) + 96 weeks (Part B)
Incidence of neutralizing antibodies against empasiprubart in serum | up to 24 weeks (Part A) + 96 weeks (Part B)
Incidence of (serious) adverse events | up to 24 weeks (Part A) + 96 weeks (Part B)
Percentage change from baseline in free C2 and total C2 over time | up to 24 weeks (Part A) + 96 weeks (Part B)
Serum concentrations of empasiprubart over time | up to 24 weeks (Part A) + 96 weeks (Part B)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (9):
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Homestead Associates in Research Inc, Homestead, Florida
  - Visionary Investigators Network, Miami, Florida
  - Paradigm Health System, Slidell, Louisiana
  - Erlanger Health System, Columbia, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - NeuroCarePlus, Houston, Texas
  - National Neuromuscular Research Institute, Irving, Texas
- Estonia (2):
  - Astra Kliinik, Tallinn
  - Tartu University Hospital, Tartu
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Japan (3):
  - Chiba University Hospital, Chūōku
  - Osaka Metropolitan University Hospital, Osaka
  - General Hospital Tsuchiura Kyodo Hospital, Tsuchiura
- Poland (4):
  - Neurocentrum Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Neurologia Slaska, Katowice
  - Centrum Medyczne Linden, Krakow
  - Centrum Medyczne Medyk, Rzeszów
- ULS de Santo António, EPE - Hospital de Santo António, Porto, Portugal
- Institutul National de Neurologie si Boli Neurovasculare Bucuresti, Bucharest, Romania
- Univerzitna nemocnica MARTIN, Martin, Slovakia
- South Korea (3):
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Hospital Universitario Vall d'Hebron, Sant Andreu de la Barca, Spain
- Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No